CLINICAL TRIAL: NCT04672590
Title: COVID-19 Neurological Disease: A Prospective Study in Brazil, India and Malawi
Brief Title: COVID-19 Neurological Disease: A Prospective Study
Status: Completed | Type: Observational
Sponsor: University of Liverpool (Other)
Collaborators: Christian Medical College, Vellore, India (Other); Instituto Autoimune, Brazil (Unknown); University College London Hospitals (Other); Oswaldo Cruz Foundation (Other); Kamuzu University of Health Sciences (Other); National Institute of Mental Health and Neuro Sciences, India (Other); Encephalitis Society, UK (Unknown)
Responsible Party: Sponsor
Other Study IDs: UoL001596
Record Dates: First submitted 2020-12-09; First posted 2020-12-17 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Diseases of the Nervous System; Other Specified Viral Diseases
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cases: Patients admitted to a study hospital meeting criteria for confirmed or probable acute new-onset neurological disease and confirmed or probable COVID-19.
  Interventions: Other: Primary exposure is hypoxia (no intervention)
- Controls: Patients admitted to a study hospital meeting criteria for confirmed or probable COVID-19, without confirmed or probable acute new-onset neurological disease.
  Interventions: Other: Primary exposure is hypoxia (no intervention)

INTERVENTIONS:
Other: Primary exposure is hypoxia (no intervention) — The primary exposure, hypoxia, will be defined as severe, non-severe or none for each participant, based on pre-defined criteria.

SUMMARY:
Background: Recent reports increasingly recognize neurological manifestations in COVID-19 patients. However, the full spectrum of the disease and risk factors are not well understood.

Aim: To describe the full spectrum of neurological manifestations in COVID-19 and assess the clinical characteristics, risks and prognostic factors.

Outcomes: Identification of COVID-19 associated neurological disease is the primary outcome while requirement for admission to critical care unit, mortality, length of hospital stay, quality of life, and neurological disability are the secondary outcomes.

Participants: Patients above Age more than 18 years enrolled based on new-onset acute neurological disease and COVID19 positive will serve as cases while patient with confirmed COVID-19 without neurological manifestation will serve as controls.

Design and Procedures: The study is prospective case control in design and is divided into three phases in India, Brazil and Malawi ; the first phase will address role of hypoxia in causation of neurological diseases, the second phase will compare characteristics of patients hospitalized with COVID-19 with and without neurological disease and the third phase will assess the long-term follow up (at 3 months and 9 months) of cases.

ELIGIBILITY:
Cases

Inclusion criteria:

1. Confirmed or probable new-onset acute neurological disease (according to study definitions) AND
2. Confirmed or probable COVID-19 (according to study definitions), diagnosed using tests performed no later than 5 days after presentation with neurological disease

Exclusion criteria (any of):

* Age <18 years
* Neurological features are explained fully by a previous neurological disease
* PCR test performed >5 days after admission to hospital, in the absence of clinical illness meeting criteria for suspected COVID-19 (to exclude those with hospital-acquired infection).
* Enrolled on the basis of new-onset acute neurological disease, but subsequently does not meet definition for probable or confirmed COVID-19.

Controls

Two controls with non-neurological COVID-19 will be recruited per case.

They will meet all of the following criteria:

* Adults, no more than 5 years younger or older than the case.
* Enrolled at a similar time since admission to hospital as the case, defined as: <7 days; 7-13 days inclusive; or ≥14 days.
* Hospitalised patients with confirmed or probable COVID-19 (according to study definitions)
* Not meeting criteria for confirmed or probable new-onset acute neurological disease (according to study definitions).

Some potential controls may be reclassified as cases if they develop neurological manifestations at up to 30 days after admission to hospital.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases: Hospitalised patients with acute new-onset neurological disease and COVID-19
  Controls: Hospitalised patients with COVID-19, without acute new-onset neurological disease
Sampling Method: Non-Probability Sample
Enrollment: 1017 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Acute new-onset neurological disease | Day 30 of admission, or at discharge, or at death, whichever is earlier

SECONDARY OUTCOMES:
Admission to a critical (intensive/high dependency) care unit | Day 30 of admission, or at discharge, or at death, whichever is earlier
Time to discharge from hospital | Day 30 of admission, or at discharge, or at death, whichever is earlier
Severity of stroke using National Institutes of Health Stroke Scale (NIHSS) | Day 30 of admission, or at discharge, or at death, whichever is earlier
  A score made up of 11 elements. Total min 0; max 42. Lower is better; 0 can be scored if the person has full function in every element of the assessment.
Glasgow Outcome Scale Extended | Discharge (or day 30), 3 months and 9 months
  An ordinal scale, from 1 = death (minimum; worst outcome) to 8 = upper good recovery (maximum; best outcome).
Modified Rankin Score | Discharge (or day 30), 3 months and 9 months
  Modified Rankin Score using a simplified algorithm by Bruno et al 2010. An ordinal scale, from 0 = no symptoms at all (minimum; best outcome) to 6 = dead (maximum; worst outcome).
Montreal Cognitive Assessment (MoCA) | Discharge (or day 30), 3 months and 9 months
  Montreal Cognitive Assessment (MoCA), using a full test at discharge (or day 30) and a telephone test at 3 months and 9 months
Development of new onset neurological sequelae | Discharge (or day 30), 3 months and 9 months
  Development of new onset neurological sequelae e.g.epilepsy, new/recurrent stroke, cognitive decline, encephalitis
European QoL-5D (EQ-5D-3L) overall health utility quality of life score | Discharge (or day 30), 3 months and 9 months
  A questionnaire scoring 5 domains of quality of life at ordinal levels of 1-3 each (1 = best; 3 = worst), plus an overall health state score from 0 to 100 on a visual analog scale (0 = worst; 100 = best).
Death | In-hospital (up to 30 days from admission), and at 3 months and 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Tom Solomon, PhD, Principal Investigator — University of Liverpool
Locations (5):
- FioCruz, Recife, Brazil
- India (2):
  - National Institute of Mental Health and Neurosciences, Bangalore
  - Christian Medical College, Vellore
- Malawi (2):
  - Malawi Liverpool Wellcome Clinical Research Programme, Blantyre
  - Kamuzu University of Health Sciences, Blantyre

IPD SHARING:
Plan to Share IPD: Yes
Limited dataset